CLINICAL TRIAL: NCT03719157
Title: Comparison of OSTAP, ESP Block,Injection of Local Anesthetic to Trocar Insertion for Elective Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Burak Nalbant, Assistant Doctor, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain; Regional Anesthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Unilateral ESP Block (Active Comparator): Before general anaesthesia, Ultrasound guided unilateral ESP block will perform with 15 ml of 0.5% bupivacaine and 5 ml 2% lidocaine.Patient controlled analgesia (PCA) with tramadol will apply to the all patients. Postoperative pain assessment and opioid consumption will record till the postoperative 24 th hours.
  Interventions: Procedure: Unilateral ESP Block; Drug: intravenous patient controlled analgesia
- Unilateral OSTAP block (Active Comparator): Under general anaesthesia, Ultrasound guided unilateral OSTAP block will perform with 15 ml of 0.5% bupivacaine and 5 ml 2% lidocaine.Patient controlled analgesia (PCA) with tramadol will apply to the all patients. Postoperative pain assessment and opioid consumption will record till the postoperative 24 th hours.
  Interventions: Procedure: Unilateral OSTAP Block; Drug: intravenous patient controlled analgesia
- Injection of Local Anesthetic to Trocar Insertion (Active Comparator): After the laparoscopic surgery was completed, the trocar incision sites were closed. Following the infiltration rules, local anesthetic (15 ml of 0.5% bupivacaine and 5 ml 2% lidocaine) was applied to the trocar sites of skin, fascia, muscle, and preperitoneal area by the surgical team after the operation. A total of 20 mL of local anesthetic was used, with 6 mL for trocar sites of 10 mm, and 4 mL for trocar sites of 5 mm .Patient controlled analgesia (PCA) with tramadol will apply to the all patients. Postoperative pain assessment and opioid consumption will record till the postoperative 24 th hours.
  Interventions: Procedure: Injection of Local Anesthetic to Trocar Insertion; Drug: intravenous patient controlled analgesia
- multimodal analgesia (Sham Comparator): Perioperative and postoperative routine analgesic protocol will be performed with no additional regional anesthesia method.Patient controlled analgesia (PCA) with tramadol will apply to the all patients. Postoperative pain assessment and opioid consumption will record till the postoperative 24 th hours.
  Interventions: Drug: intravenous patient controlled analgesia

INTERVENTIONS:
Procedure: Unilateral ESP Block — USG guided ESP block will perform unilateral with Bupivacaine and Lidocain mixture
  Arms: Unilateral ESP Block
Procedure: Unilateral OSTAP Block — USG guided OSTAP block will perform unilateral with Bupivacaine and Lidocain mixture
  Arms: Unilateral OSTAP block
Procedure: Injection of Local Anesthetic to Trocar Insertion — Bupivacaine infiltration will be performed at the end of the surgical procedure to trocar insertion sites.
  Arms: Injection of Local Anesthetic to Trocar Insertion
Drug: intravenous patient controlled analgesia — All patients were followed using a standardized postoperative analgesia protocol which includes tramadol PCA. Tramadol at a concentration of 5 mg/mL is included in our PCA protocol (total volume 100 mL.) PCAs were set to no basal infusion and 10 mg bolus doses with a 20 min lock time.

SUMMARY:
Main purpose of this prospective single center randomized study is to compare the analgesic effect of ultrasound guided Unilateral Oblique Subcostal Transversus Abdominis Plane (TAP),unilateral Erector Spinae Plane (ESP) blocks and Port site infiltration of local anesthetic in subjects undergoing laparoscopic cholecystectomy. Total 100 patients, American society of anaesthesiology physical status I-II aged between 18-65 who underwent laparoscopic cholecystectomy will recruit to the study.

ELIGIBILITY:
Inclusion Criteria:

* ASA Status 1-2 patients Exclusion criteria
* Patients with a body mass index (BMI) of >40kg/m2
* ASA score of >III
* Previous abdominal surgery
* Pregnant or breastfeeding patients
* Patients with coagulopathy
* Known local anesthetic allergy
* infection at the injection site

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 24 hours
  Patient controlled analgesia (PCA) will provide with tramadol PCA. Total tramadol consumption will calculate and record till the postoperative 24th hours.
Postoperative pain scores: NRS | 24 hours
  Postoperative pain assessment will apply with numerical rating scale. These scores will record till the postoperative 24 th hours.

SECONDARY OUTCOMES:
postoperative nause and vomiting | 24 hours
  The patient with nausea and vomiting will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Diskapi education and research hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nalbant B, Donmez A, Altinsoy S, Kavak Akelma F. Efficacy of OSTAP, ESP block, trocar site local anesthetic injection in elective laparoscopic cholecystectomy: A randomized controlled trial. Medicine (Baltimore). 2025 Aug 1;104(31):e43607. doi: 10.1097/MD.0000000000043607. PMID 40760576